CLINICAL TRIAL: NCT06005350
Title: Validation of an Enzymatic Assay for Quantification of Nicotinamide Adenine Dinucleotide in Blood Plasma After Ingestion of the Vitamin B3 Variant Nicotinamide Riboside: a Randomized Controlled Trial
Brief Title: Nicotinamide Riboside Impact on Extracellular Nicotinamide Adenine Dinucleotide (NAD+)
Acronym: NICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Principal Investigator, Felix Krenzien, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EA4/210/19
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: NAD
Keywords: Nicotinamide riboside; extracellular NAD+; enzymatic assay
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NR-Treatment (Experimental): NR-Chloride Preparation 1000mg/day for 10 days
  (500mg - 0 - 500mg -0)
  Interventions: Dietary Supplement: Niagen
- Placebo (Placebo Comparator): Placebo for 10 days
  (1 - 0 - 1 - 0)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Niagen — Nicotinamide-Riboside-Chloride Preparation 1000mg/day
  Arms: NR-Treatment
Other: Placebo — Placebo Preperation
  Arms: Placebo

SUMMARY:
The investigation is a clinical study in which the impact of taking the dietary supplement nicotinamide riboside (NR) on the concentration of extracellular nicotinamide adenine dinucleotide (eNAD+) in human plasma over time will be determined. The study will be conducted in a randomized, double-blinded, and placebo-controlled manner.

DETAILED DESCRIPTION:
The significance of nicotinamide adenine dinucleotide (NAD+) in promoting a healthy life is currently under intense research. Despite an increasing number of research groups focusing on NAD+, there is no validated measurement method for extracellular NAD+. With this research project, the investigators aim to address this research gap.

The coenzyme NAD+ is one of the central regulators of metabolism, existing mostly in its oxidized form, NAD+, and its reduced form, NADH, in a dynamic equilibrium. NAD+ is indispensable for various metabolic processes, and is especially key in ATP generation. It also enables gluconeogenesis, ketogenesis, pentose phosphate production, heme and lipid synthesis, and the elimination of oxygen radicals.

To validate the NAD+ assay as a robust and reliable quantification method of extracellular NAD+, a controlled increase of the measured metabolite in blood plasma is required through NAD+ precursor administration.

Multiple studies have already demonstrated that oral NR intake can increase NAD+ levels in mammalian cells, rodent tissues, and peripheral blood mononuclear cells (PBMCs) in humans. However, this relationship has not been explored in the extracellular space due to the lack of reliable quantification of eNAD+ levels. Now, using the NAD+ assay, the investigators aim to examine the increase of eNAD+ after oral NR intake and provide initial data on the effects of a 1000 mg/day dosage.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Normal nutritional status and
* Age >18 years.

Exclusion Criteria:

* Pregnancy and/or lactation, or
* Severe psychiatric disorders, or
* Conditions that involve attention deficits, or
* Severe medical conditions, or
* Withdrawal of consent by the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
NR increases plasma concentrations of eNAD+ | 10 days
  The daily intake of 1,000 mg of NR changes the concentration of eNAD+ over the course of 10 days. The NAD+ assay measures the changes in concentrations of eNAD+ in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Clinic, Campus Virchow-Klinikum / Campus Charité Mitte, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogan KL, Brenner C. Nicotinic acid, nicotinamide, and nicotinamide riboside: a molecular evaluation of NAD+ precursor vitamins in human nutrition. Annu Rev Nutr. 2008;28:115-30. doi: 10.1146/annurev.nutr.28.061807.155443. PMID 18429699
- [Background] Brunnbauer P, Leder A, Kamali C, Kamali K, Keshi E, Splith K, Wabitsch S, Haber P, Atanasov G, Feldbrugge L, Sauer IM, Pratschke J, Schmelzle M, Krenzien F. The nanomolar sensing of nicotinamide adenine dinucleotide in human plasma using a cycling assay in albumin modified simulated body fluids. Sci Rep. 2018 Oct 31;8(1):16110. doi: 10.1038/s41598-018-34350-6. PMID 30382125
- [Background] Canto C, Houtkooper RH, Pirinen E, Youn DY, Oosterveer MH, Cen Y, Fernandez-Marcos PJ, Yamamoto H, Andreux PA, Cettour-Rose P, Gademann K, Rinsch C, Schoonjans K, Sauve AA, Auwerx J. The NAD(+) precursor nicotinamide riboside enhances oxidative metabolism and protects against high-fat diet-induced obesity. Cell Metab. 2012 Jun 6;15(6):838-47. doi: 10.1016/j.cmet.2012.04.022. PMID 22682224
- [Background] Chi Y, Sauve AA. Nicotinamide riboside, a trace nutrient in foods, is a vitamin B3 with effects on energy metabolism and neuroprotection. Curr Opin Clin Nutr Metab Care. 2013 Nov;16(6):657-61. doi: 10.1097/MCO.0b013e32836510c0. PMID 24071780
- [Background] Dolopikou CF, Kourtzidis IA, Margaritelis NV, Vrabas IS, Koidou I, Kyparos A, Theodorou AA, Paschalis V, Nikolaidis MG. Acute nicotinamide riboside supplementation improves redox homeostasis and exercise performance in old individuals: a double-blind cross-over study. Eur J Nutr. 2020 Mar;59(2):505-515. doi: 10.1007/s00394-019-01919-4. Epub 2019 Feb 6. PMID 30725213
- [Background] Imai SI, Guarente L. It takes two to tango: NAD+ and sirtuins in aging/longevity control. NPJ Aging Mech Dis. 2016 Aug 18;2:16017. doi: 10.1038/npjamd.2016.17. eCollection 2016. PMID 28721271
- [Background] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Background] Yoshino J, Baur JA, Imai SI. NAD+ Intermediates: The Biology and Therapeutic Potential of NMN and NR. Cell Metab. 2018 Mar 6;27(3):513-528. doi: 10.1016/j.cmet.2017.11.002. Epub 2017 Dec 14. PMID 29249689